CLINICAL TRIAL: NCT02957799
Title: A Randomized Controlled Trial to Improve the South African Government's Community Health Workers' Capacities to Deliver Evidence-based Interventions for Optimizing HIV Outcomes and Reducing Its Comorbidities
Brief Title: Improving South African Government Workers' Capacities to Deliver HIV Interventions
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of Stellenbosch (Other)
Responsible Party: Principal Investigator, Mary Jane Rotheram-Borus, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01MH111391 (NIH); R01MH111391 (NIH)
Record Dates: First submitted 2016-10-26; First posted 2016-11-08 (Estimated); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: HIV; Partner Violence; Malnutrition; Alcohol Use/Abuse; Depression
Keywords: Pregnancy; Home Healthcare Visits; Community Health Workers; Infants
MeSH Terms: conditions — Malnutrition; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Accountable Condition- 8 clinics (Experimental): In the Accountable Condition, the intervention includes mothers who will receive home visits from government-funded CHW who will be trained once under Philani and receive ongoing monitoring and supervision.
  Interventions: Behavioral: Accountable Condition
- Control Condition- 8 clinics (Experimental): The Control Condition will include mothers who receive home visits from government-funded CHW who will be trained once under Philani and receive supervision and monitoring consistent with local government practices.
  Interventions: Behavioral: Control Condition

INTERVENTIONS:
Behavioral: Accountable Condition — Mothers will receive home visits by government-funded CHW who will be trained under Philani as well as receive ongoing monitoring and supervision. CHW will monitor mother's health and linkage to care; CHW will refer all mothers to local clinics for HIV, blood sugar, and pregnancy testing. CHW will also have a mobile phone to record information at each visit. CHW will log their home visits each day, rate the content and skills addressed on the mobile phone, weigh children, and report outcome achievements (e.g., receiving the child grant, immunizations, breastfeeding, and retention/ adherence to HIV care). The CHW in this arm will receive data-informed supervision. CHW will be monitored weekly with review of contact logs, recorded outcomes, and random site visits by supervising in-service training on a monthly basis. The Accountable Condition will last for two years (until the child is 24 months old).
  Arms: Accountable Condition- 8 clinics
Behavioral: Control Condition — Mothers will receive home visits by government-funded CHW who will be trained under Philani as well as receive supervision and monitoring consistent with local government practices. CHW will monitor mother's health and linkage to care. CHW will refer all mothers to local clinics for HIV, blood sugar, and pregnancy testing. The Control Condition will last for two years (until the child is 24 months old).
  Arms: Control Condition- 8 clinics

SUMMARY:
The purpose of this study is to address the United States Office of AIDS Research highest priorities: improving the workforce, reducing health disparities, and addressing HIV comorbidities. UCLA will randomize the government-funded community health workers (CHW) from 16 clinics in matched rural areas in the Eastern Cape in South Africa to either: 1) the Accountable Condition (AC) in which additional monitoring and accountability systems that Philani routinely uses are implemented or 2) a Control Condition (CC), of initial Philani training, but ongoing supervision and monitoring consistent with local government practices.

DETAILED DESCRIPTION:
Each dollar invested in maternal, child health (MCH) yields a nine-fold benefit. Home visiting has been repeatedly demonstrated efficacious in improving MCH outcomes, including when delivered by CHW in low and middle income countries (LMIC). However, when home visiting programs are scaled, they are not effective. Africa has particular challenges with broad implementation of effective interventions often associated with the poorly trained and poorly monitored health personnel, in this case, CHW who are perinatal home visitors.

The investigators have shown that with training, supervision, and accountability, CHW home visits are effective in a successful randomized controlled trial (RCT) conducted in peri-urban townships in Cape Town, South Africa. CHW were trained to address HIV, alcohol, and malnutrition among all pregnant women in a neighborhood - to avoid stigma and to address multiple challenges concurrently. The visits significantly improved maternal and child outcomes over three years. Based on these results, the Philani Intervention Model served as one model for re-engineering primary health care for 65,000 CHW in South Africa. The Mthatha Provincial Government has agreed for the Philani Program to train, monitor, and supervise their already-hired CHW. This RCT will evaluate whether routinely implementing training and monitoring CHW behavior and MCH outcomes with mobile phones, and providing data-informed supervision, will result in CHW becoming more effective. Stellenbosch University interviewers will independently assess outcomes of each mother at pregnancy, and of the mothers and infants within two weeks of post-birth, 6 months, 15 months, and 24 months later. The primary outcome will be maternal HIV/TB testing, linkage to care, treatment adherence and retention in medical regimens, depression, and parenting; and her child's physical growth, cognitive functioning, and behavior adjustment.

ELIGIBILITY:
Inclusion Criteria:

* Mothers living in the catchment area
* Mothers not identified as psychotic or delusional based on the interviewer's judgment
* Mothers able to provide informed consent

Exclusion Criteria:

* Inability to give informed consent
* Inability to converse with the interviewer or the CHW
* Death of the mother or infant.

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 840 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Number of significantly improved child and maternal outcomes | 2 Years
  Out of 10 variables, the investigators total number of outcomes that are significantly better in the Accountable Condition compared to the Control Condition. The variables are for mothers and children:
  For Mothers:
  1. Adhere to medical regimens
  2. Breastfeed for six months (mixed ok)
  3. No alcohol after learning that the participant was pregnant
  4. Mental health, EPDS
     For Children:
  5. Growth in height (<-2SD)
  6. Growth in weight (<-2SD)
  7. Number of Hospitalizations
  8. WHO developmental scale measure in normal range
  9. In normal range of CBCL
  10. In normal range on the Bayley

SECONDARY OUTCOMES:
Number of significantly improved child and maternal outcomes for HIV positive mothers | 2 Years
  Out of 9 variables, the investigators total the number of outcomes that are significantly better in the Accountable Condition compared to the Control Condition for HIV positive mothers. The variables are:
  1. ARV 6 weeks before birth
  2. NVP at birth
  3. Cipro for child
  4. TB testing
  5. AZT for child
  6. PCR testing at 6 weeks
  7. Get the results of PCR testing
  8. One feeding method for 6 months
  9. Breastfeed solely for 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Jane Rotheram-Borus, Principal Investigator — Study Principal Investigator Department of Psychiatry & Biobehavioral Sciences, Semel Institute, UCLA
Locations (2):
- South Africa (2):
  - Stellenbosch University, Stellenbosch
  - Zithulele Hospital, Zithulele

IPD SHARING:
Plan to Share IPD: Yes
At the conclusion of this study we have a plan to de-identify the data and to make it available to other researchers.

REFERENCES:
- [Derived] Minozzi S, Ambrosi L, Saulle R, Uhm SS, Terplan M, Sinclair JM, Agabio R. Psychosocial and medication interventions to stop or reduce alcohol consumption during pregnancy. Cochrane Database Syst Rev. 2024 Apr 29;4(4):CD015042. doi: 10.1002/14651858.CD015042.pub2. PMID 38682758
- [Derived] Rotheram-Borus MJ, le Roux KW, Norwood P, Stansert Katzen L, Snyman A, le Roux I, Dippenaar E, Tomlinson M. The effect of supervision on community health workers' effectiveness with households in rural South Africa: A cluster randomized controlled trial. PLoS Med. 2023 Mar 2;20(3):e1004170. doi: 10.1371/journal.pmed.1004170. eCollection 2023 Mar. PMID 36862754
- [Derived] Rotheram-Borus MJ, Le Roux K, Le Roux IM, Christodoulou J, Laurenzi C, Mbewu N, Tomlinson M. To evaluate if increased supervision and support of South African Government health workers' home visits improves maternal and child outcomes: study protocol for a randomized control trial. Trials. 2017 Aug 7;18(1):368. doi: 10.1186/s13063-017-2074-5. PMID 28784142